CLINICAL TRIAL: NCT04213131
Title: Efficacy and Safety of hUC-MSCs and hUCB-MSCs in the Treatment of Chronic Spinal Cord Injury: a Prospective, Randomized, Open-label, Parallel, and Controlled Clinical Study
Brief Title: Efficacy and Safety of hUC-MSCs and hUCB-MSCs in the Treatment of Chronic Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Liu Jing, Chief Physician, The First Affiliated Hospital of Dalian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstHospitalDalianMU005
Record Dates: First submitted 2019-12-20; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Cord Blood Stem Cell Transplantation; Pain; Human
MeSH Terms: conditions — Spinal Cord Injuries; Pain | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: participants are assigned to one of two or more groups in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Rehabilitation control group (Other): Routine rehabilitation treatment for chronic spinal cord injury and Intravenous injection of 100 mL 0.9% saline solution.
  Interventions: Other: Stem cell transplantation
- hUC-MSCs intravenous administration group (Experimental): intravenous administration of 100 mL of cell suspension containing 5×107 hUC-MSCs
  Interventions: Other: Stem cell transplantation
- hUC-MSCs lumbar administration group (Experimental): lumbar administration of a solution prepared by 5 mL of cell suspension containing 5×107 hUC-MSCs and 5 mL of cerebrospinal fluid
  Interventions: Other: Stem cell transplantation
- hUC-MSCs local administration group (Experimental): hUC-MSCs (100,000 cells/μL) were injected via 4 points in the edge of injured spinal cord (2 points in the upper edge and 2 points in the lower edge), 16 μL hUC-MSCs/point.
  Interventions: Other: Stem cell transplantation
- hUCB-MSCs intravenous administration group (Experimental): intravenous administration of 100 mL of cell suspension containing 5×107 hUCB-MSCs
  Interventions: Other: Stem cell transplantation
- hUCB-MSCs lumbar administration group (Experimental): lumbar administration of a solution prepared by 5 mL of cell suspension containing 5×107 hUCB-MSCs and 5 mL of cerebrospinal fluid
  Interventions: Other: Stem cell transplantation
- hUCB-MSCs local administration group (Experimental): hUCB-MSCs (100,000 cells/μL) were injected via 4 points in the edge of injured spinal cord (2 points in the upper edge and 2 points in the lower edge), 16 μL hUCB-MSCs/point.
  Interventions: Other: Stem cell transplantation

INTERVENTIONS:
Other: Stem cell transplantation — The eligible patients with chronic spinal cord injury included in this study will receive intravenous, lumbar, and local administration of hUC-MSCs/hUCB-MSCs and routine rehabilitation treatment. At 1, 3, 6 and 12 months after treatment, patients will be followed up and evaluated.

SUMMARY:
There is evidence that human umbilical cord blood-derived mesenchymal stem cells (hUCB-MSCs) can differentiate into oligodendrocytes and neurons, and improve the recovery of nerve function, which strongly suggests the feasibility and effectiveness of hUCB-MSCs as an intervention treatment for spinal cord injury. At present, there are only a few clinical centers in which hUCB-MSCs transplantation for treatment of chronic spinal cord injury has been performed and a certain degree of efficacy has been achieved. However, this has not been supported by systematic standardized randomized controlled trials. Therefore, the investigators design a prospective, randomized, open-label, parallel, controlled trial to evaluate the efficacy of human umbilical cord-derived mesenchymal stem cells (hUC-MSCs)/hUCB-MSCs to treat spinal cord injury. The primary objective of this study was to investigate whether hUC-MSCs)/hUCB-MSCs transplantation can improve the locomotor function of patients with spinal cord injury. The secondary objectives were to investigate whether hUC-MSCs)/hUCB-MSCs transplantation can improve the muscle tension of patients with spinal cord injury and investigate the complications and safety of hUC-MSCs)/hUCB-MSCs transplantation.

DETAILED DESCRIPTION:
Patient recruitment will be performed via information dissemination on bulletin boards to advertise the study among patients at the clinics and wards of the First Affiliated Hospital of Dalian Medical University, China. Patients interested in participation in this study or their legal guardians contact the project manager via telephone. Patients will be screened according to the inclusion and exclusion criteria after providing signed informed consent. Eligible patients with chronic spinal cord injury will receive intravenous, lumbar, and local administration of hUC-MSCs/hUCB-MSCs (provided by Cell Bank of Stem Cell Clinical Research Institute, The First Affiliated Hospital of Dalian Medical University). The primary outcome measure of this study is neurologic function scores, including ASIA (American Spinal Injury Association) motor score, ASIA sensory score, ASIA impairment scale (ASIA classification), and acupuncture score. These scores will be used to evaluate the recovery of nerve function after spinal cord injury and determine the therapeutic efficacy and persistence. The secondary outcome measures of this study include Walking Index of Spinal Cord Injury (WISCI), Spinal Cord Independence Measure (SCIM), Kunming Locomotion Scale (KLS), Modified Ashworth Scale (MAS), and Visual Analogous Scale (VAS) scores and the incidence of adverse reactions. At 1, 3, 6 and 12 months after treatment, patients will be followed up to evaluate the efficacy and safety of hUC-MSCs)/hUCB-MSCs transplantation in the treatment of spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age at 20-65 years, of either gender;
* Patients with radiologically confirmed chronic spinal cord injury, with over 1 year of disease history;
* Patients having no change in ASIA motor score, ASIA sensory score, ASIA impairment scale (ASIA classification) score, and acupuncture score within 6 months and no change in recovery of neurological function;
* Patients with spinal cord injury who have been relieved of spinal cord compression injury or hematoma clearance;
* Patients with trauma-caused spinal cord injury accompanied by neurological deficits (sensory, motor, and autonomic dysfunction);
* Patients who have been subjected to electromyography and urodynamics examination to determine the denervation below the level of spinal cord injury and the function of the detrusor muscle;
* Patients with normal results of routine blood, urine, and stool tests, blood biochemical parameters, coagulation function, immune indices, electrocardiography and chest radiograph findings, and negative results of human immunodeficiency viruses and syphilis antibody
* Provision of written informed consent; approval by hospital ethics committee

Exclusion Criteria:

* Patients with consciousness disorder, lumbosacral infection, or other complications;
* Patients with spinal cord injury caused by spinal cord compression, syringomyelia, subacute combined degeneration of spinal cord, spinal vascular disease, arachnoiditis of spinal cord, radiation myelopathy, amyotrophic lateral sclerosis, multiple sclerosis, or neuromyelitis optica;
* Patients with cerebrovascular disease, peripheral neuropathy, history of epilepsy, pregnancy, lactation, diabetes mellitus, mental disorders or other factors that affect the clinical treatment of spinal cord injury;
* Patients with serious cardiopulmonary disease, liver and kidney function damage, and other serious basic diseases;
* Patients wearing a metal internal fixator (except titanium alloy) or a pacemaker in the body;
* Patients with poor compliance who are unable to complete the study process or who are not considered suitable for the study by the investigators;
* Decline to participate in this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Neurologic function score | Change from Baseline at 12 months after treatment
  ASIA motor score, ASIA sensory score, ASIA impairment scale (ASIA classification), and acupuncture score will be obtained to evaluate the recovery of nerve function after spinal cord injury and determine the therapeutic efficacy and persistence.

SECONDARY OUTCOMES:
Walking Index of Spinal Cord Injury (WISCI) | Change from Baseline at 12 months after treatment
  To evaluate walking ability
Spinal Cord Independence Measure (SCIM) | Change from Baseline at 12 months after treatment
  To evaluate ability of daily activities after spinal cord injury
Kunming Locomotion Scale (KLS) | Change from Baseline at 12 months after treatment
  To evaluate walking ability
Modified Ashworth Scale (MAS) | Change from Baseline at 12 months after treatment
  0-4 score, to evaluate spasticity
Visual Analogous Scale (VAS) | Change from Baseline at 12 months after treatment
  To evaluate the degree of pain

OTHER OUTCOMES:
Incidence of adverse reactions | Before and 1, 3, 6, and 12 months after treatment
  To record adverse reactions after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Ph.D, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China